CLINICAL TRIAL: NCT04560374
Title: The Effect of Using Crochet Octopus in Reducing The Pain Developed During The Process of Heel Lance İn Neonates: A Randomized Controlled Study
Brief Title: Crochet Octopus in The Process of Heel Lance in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, cagri covener ozcelik, Associate Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 90139838-000-E.20252
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Procedural Pain
Keywords: neonate; pain; heel lance; developmental care
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Crochet octopus was delivered to the hands of the neonates in the experimental group 10 minutes before heel lance process and they were contacted with the crochet octopus up to 10 minutes after the procedure.
  Interventions: Device: crochet octopus
- Control Group (No Intervention): Control group neonates were performed all the process without delivering them any crochet octopus.

INTERVENTIONS:
Device: crochet octopus — Delivering crochet octopus to the hands of the neonates
  Arms: Experimental Group

SUMMARY:
The main objective of the study was to determine the effect of using crochet octopus in order to reduce the acute pain developed during the process of heel lance in neonates.

The hypothesis of the study was "Crochet octopus is rather effective in reducing the acute pain in heel lance process for neonates".

DETAILED DESCRIPTION:
The study was conducted as randomized controlled. It included term neonates born between May 2020 and August 2020 at a training and research hospital. The study was completed with 100 neonates in total as 50 for experiment and 50 for control groups. During the process of heel lance, experiment group neonates were delivered crochet octopus 10 minutes before the process and let them touch the octopus 10 minutes more after the process. Control group neonates experienced the process without any intervention. As for the data collection, "Newborn Identification Form", "Neonatal-Infant Pain Scale (NIPS)" and "Observation Form" were utilized. The whole process was video-recorded.

ELIGIBILITY:
Inclusion Criteria:

* being a healthy term neonates,
* being 5-15 days,
* taking of blood sample for Guthrie test routinely.

Exclusion Criteria:

* admitted to the neonatal intensive care units
* his/her being taken any analgesics prior to the intervention,
* having any congenital anomalies

Ages: 5 Days to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cagri Covener Ozcelik, PhD, Study Chair — Marmara University; Özge Eren, MSN, Principal Investigator — Marmara University; Nagihan Sabaz, MSN, Principal Investigator — Marmara University; Muhammet Bulut, MD, Principal Investigator — Giresun University
Locations (1):
- Giresun University Women and Children's Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasoglu A, Cabioglu MT, Tugcu AU, Ince DA, Tekindal MA, Ecevit A, Tarcan A. Acupressure at BL60 and K3 Points Before Heel Lancing in Preterm Infants. Explore (NY). 2015 Sep-Oct;11(5):363-6. doi: 10.1016/j.explore.2015.07.005. Epub 2015 Jul 3. PMID 26242287
- [Background] Akcan E, Polat S. Comparative Effect of the Smells of Amniotic Fluid, Breast Milk, and Lavender on Newborns' Pain During Heel Lance. Breastfeed Med. 2016 Aug;11(6):309-314. doi: 10.1089/bfm.2015.0174. Epub 2016 Jun 17. PMID 27315487
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn; American Academy of Pediatrics Section on Surgery; Canadian Paediatric Society Fetus and Newborn Committee; Batton DG, Barrington KJ, Wallman C. Prevention and management of pain in the neonate: an update. Pediatrics. 2006 Nov;118(5):2231-41. doi: 10.1542/peds.2006-2277. PMID 17079598
- [Background] Anand KJ; International Evidence-Based Group for Neonatal Pain. Consensus statement for the prevention and management of pain in the newborn. Arch Pediatr Adolesc Med. 2001 Feb;155(2):173-80. doi: 10.1001/archpedi.155.2.173. PMID 11177093
- [Background] Asmerom Y, Slater L, Boskovic DS, Bahjri K, Holden MS, Phillips R, Deming D, Ashwal S, Fayard E, Angeles DM. Oral sucrose for heel lance increases adenosine triphosphate use and oxidative stress in preterm neonates. J Pediatr. 2013 Jul;163(1):29-35.e1. doi: 10.1016/j.jpeds.2012.12.088. Epub 2013 Feb 14. PMID 23415615
- [Background] Axelin A, Salantera S, Lehtonen L. 'Facilitated tucking by parents' in pain management of preterm infants-a randomized crossover trial. Early Hum Dev. 2006 Apr;82(4):241-7. doi: 10.1016/j.earlhumdev.2005.09.012. Epub 2006 Jan 10. PMID 16410042
- [Background] Bueno M, Stevens B, de Camargo PP, Toma E, Krebs VL, Kimura AF. Breast milk and glucose for pain relief in preterm infants: a noninferiority randomized controlled trial. Pediatrics. 2012 Apr;129(4):664-70. doi: 10.1542/peds.2011-2024. Epub 2012 Mar 5. PMID 22392169
- [Background] Courtois E, Droutman S, Magny JF, Merchaoui Z, Durrmeyer X, Roussel C, Biran V, Eleni S, Vottier G, Renolleau S, Desfrere L, Castela F, Boimond N, Mellah D, Bolot P, Coursol A, Brault D, Chappuy H, Cimerman P, Anand KJ, Carbajal R. Epidemiology and neonatal pain management of heelsticks in intensive care units: EPIPPAIN 2, a prospective observational study. Int J Nurs Stud. 2016 Jul;59:79-88. doi: 10.1016/j.ijnurstu.2016.03.014. Epub 2016 Mar 30. PMID 27222453
- [Background] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Background] Grunau RE. Neonatal pain in very preterm infants: long-term effects on brain, neurodevelopment and pain reactivity. Rambam Maimonides Med J. 2013 Oct 29;4(4):e0025. doi: 10.5041/RMMJ.10132. eCollection 2013. PMID 24228168
- [Background] Hebb AL, Poulin JF, Roach SP, Zacharko RM, Drolet G. Cholecystokinin and endogenous opioid peptides: interactive influence on pain, cognition, and emotion. Prog Neuropsychopharmacol Biol Psychiatry. 2005 Dec;29(8):1225-38. doi: 10.1016/j.pnpbp.2005.08.008. Epub 2005 Oct 20. PMID 16242828
- [Background] Mangat AK, Oei JL, Chen K, Quah-Smith I, Schmolzer GM. A Review of Non-Pharmacological Treatments for Pain Management in Newborn Infants. Children (Basel). 2018 Sep 20;5(10):130. doi: 10.3390/children5100130. PMID 30241352
- [Background] Hill S, Engle S, Jorgensen J, Kralik A, Whitman K. Effects of facilitated tucking during routine care of infants born preterm. Pediatr Phys Ther. 2005 Summer;17(2):158-63. doi: 10.1097/01.pep.0000163097.38957.ec. PMID 16357666
- [Background] Huang CM, Tung WS, Kuo LL, Ying-Ju C. Comparison of pain responses of premature infants to the heelstick between containment and swaddling. J Nurs Res. 2004 Mar;12(1):31-40. doi: 10.1097/01.jnr.0000387486.78685.c5. PMID 15136961
- [Background] Hall RW, Anand KJ. Pain management in newborns. Clin Perinatol. 2014 Dec;41(4):895-924. doi: 10.1016/j.clp.2014.08.010. Epub 2014 Oct 7. PMID 25459780
- [Background] Hwang MJ, Seol GH. Cerebral Oxygenation and Pain of Heel Blood Sampling Using Manual and Automatic Lancets in Premature Infants. J Perinat Neonatal Nurs. 2015 Oct-Dec;29(4):356-62. doi: 10.1097/JPN.0000000000000138. PMID 26505850
- [Background] Jain S, Kumar P, McMillan DD. Prior leg massage decreases pain responses to heel stick in preterm babies. J Paediatr Child Health. 2006 Sep;42(9):505-8. doi: 10.1111/j.1440-1754.2006.00912.x. PMID 16925535
- [Background] Johnson AN. Kangaroo holding beyond the NICU. Pediatr Nurs. 2005 Jan-Feb;31(1):53-6. PMID 15794326
- [Background] Johnston CC, Filion F, Campbell-Yeo M, Goulet C, Bell L, McNaughton K, Byron J, Aita M, Finley GA, Walker CD. Kangaroo mother care diminishes pain from heel lance in very preterm neonates: a crossover trial. BMC Pediatr. 2008 Apr 24;8:13. doi: 10.1186/1471-2431-8-13. PMID 18435837
- [Background] Johnston CC, Stevens B, Pinelli J, Gibbins S, Filion F, Jack A, Steele S, Boyer K, Veilleux A. Kangaroo care is effective in diminishing pain response in preterm neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1084-8. doi: 10.1001/archpedi.157.11.1084. PMID 14609899
- [Background] Johnston C, Campbell-Yeo M, Fernandes A, Inglis D, Streiner D, Zee R. Skin-to-skin care for procedural pain in neonates. Cochrane Database Syst Rev. 2014 Jan 23;(1):CD008435. doi: 10.1002/14651858.CD008435.pub2. PMID 24459000
- [Background] Kahraman A, Basbakkal Z, Yalaz M, Sozmen EY. The effect of nesting positions on pain, stress and comfort during heel lance in premature infants. Pediatr Neonatol. 2018 Aug;59(4):352-359. doi: 10.1016/j.pedneo.2017.11.010. Epub 2017 Nov 13. PMID 29248383
- [Background] Kostandy RR, Ludington-Hoe SM, Cong X, Abouelfettoh A, Bronson C, Stankus A, Jarrell JR. Kangaroo Care (skin contact) reduces crying response to pain in preterm neonates: pilot results. Pain Manag Nurs. 2008 Jun;9(2):55-65. doi: 10.1016/j.pmn.2007.11.004. PMID 18513662
- [Background] Kucukoglu S, Kurt S, Aytekin A. The effect of the facilitated tucking position in reducing vaccination-induced pain in newborns. Ital J Pediatr. 2015 Aug 21;41:61. doi: 10.1186/s13052-015-0168-9. PMID 26293573
- [Background] Liu M, Zhao L, Li XF. Effect of skin contact between mother and child in pain relief of full-term newborns during heel blood collection. Clin Exp Obstet Gynecol. 2015;42(3):304-8. PMID 26151998
- [Background] Livingston K, Beider S, Kant AJ, Gallardo CC, Joseph MH, Gold JI. Touch and massage for medically fragile infants. Evid Based Complement Alternat Med. 2009 Dec;6(4):473-82. doi: 10.1093/ecam/nem076. Epub 2007 Aug 6. PMID 18955228
- [Background] Losacco V, Cuttini M, Greisen G, Haumont D, Pallas-Alonso CR, Pierrat V, Warren I, Smit BJ, Westrup B, Sizun J; ESF Network. Heel blood sampling in European neonatal intensive care units: compliance with pain management guidelines. Arch Dis Child Fetal Neonatal Ed. 2011 Jan;96(1):F65-8. doi: 10.1136/adc.2010.186429. PMID 21177753
- [Background] Meek J, Huertas A. Cochrane review: Non-nutritive sucking, kangaroo care and swaddling/facilitated tucking are observed to reduce procedural pain in infants and young children. Evid Based Nurs. 2012 Jul;15(3):84-5. doi: 10.1136/ebnurs-2011-100453. Epub 2012 Mar 12. No abstract available. PMID 22411160
- [Background] Morrow C, Hidinger A, Wilkinson-Faulk D. Reducing neonatal pain during routine heel lance procedures. MCN Am J Matern Child Nurs. 2010 Nov-Dec;35(6):346-54; quiz 354-6. doi: 10.1097/NMC.0b013e3181f4fc53. PMID 20926970
- [Background] Perry M, Tan Z, Chen J, Weidig T, Xu W, Cong XS. Neonatal Pain: Perceptions and Current Practice. Crit Care Nurs Clin North Am. 2018 Dec;30(4):549-561. doi: 10.1016/j.cnc.2018.07.013. PMID 30447813
- [Background] Pillai Riddell RR, Racine NM, Turcotte K, Uman LS, Horton RE, Din Osmun L, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Gerwitz-Stern A. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD006275. doi: 10.1002/14651858.CD006275.pub2. PMID 21975752
- [Background] Shah SR, Kadage S, Sinn J. Trial of Music, Sucrose, and Combination Therapy for Pain Relief during Heel Prick Procedures in Neonates. J Pediatr. 2017 Nov;190:153-158.e2. doi: 10.1016/j.jpeds.2017.08.003. PMID 29144240
- [Background] Smith A, Tamgumus S, Lawless S, Penrose P, EL-Khuffash A, Boyle MA. Tentacles For Tinies: The Many Arms of the Crocheted Octopus. Ir Med J. 2018 Sep 10;111(8):812. No abstract available. PMID 30415532
- [Background] Soltani S, Zohoori D, Adineh M. Comparison the Effectiveness of Breastfeeding, Oral 25% Dextrose, Kangaroo-Mother Care Method, and EMLA Cream on Pain Score Level Following Heal Pick Sampling in Newborns: a randomized clinical trial. Electron Physician. 2018 May 5;10(5):6741-6748. doi: 10.19082/6741. eCollection 2018 May. PMID 29997756
- [Background] Stevens B, Gibbins S, Franck LS. Treatment of pain in the neonatal intensive care unit. Pediatr Clin North Am. 2000 Jun;47(3):633-50. doi: 10.1016/s0031-3955(05)70230-3. PMID 10835995
- [Background] Stevens B, Yamada J, Ohlsson A, Haliburton S, Shorkey A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2016 Jul 16;7(7):CD001069. doi: 10.1002/14651858.CD001069.pub5. PMID 27420164
- [Background] Stevens B, Yamada J, Campbell-Yeo M, Gibbins S, Harrison D, Dionne K, Taddio A, McNair C, Willan A, Ballantyne M, Widger K, Sidani S, Estabrooks C, Synnes A, Squires J, Victor C, Riahi S. The minimally effective dose of sucrose for procedural pain relief in neonates: a randomized controlled trial. BMC Pediatr. 2018 Feb 23;18(1):85. doi: 10.1186/s12887-018-1026-x. PMID 29475433
- [Background] Taddio A, Katz J. The effects of early pain experience in neonates on pain responses in infancy and childhood. Paediatr Drugs. 2005;7(4):245-57. doi: 10.2165/00148581-200507040-00004. PMID 16117561
- [Background] van Sleuwen BE, L'hoir MP, Engelberts AC, Busschers WB, Westers P, Blom MA, Schulpen TW, Kuis W. Comparison of behavior modification with and without swaddling as interventions for excessive crying. J Pediatr. 2006 Oct;149(4):512-7. doi: 10.1016/j.jpeds.2006.06.068. PMID 17011324
- [Background] Whitfield MF, Grunau RE. Behavior, pain perception, and the extremely low-birth weight survivor. Clin Perinatol. 2000 Jun;27(2):363-79. doi: 10.1016/s0095-5108(05)70026-9. PMID 10863655
- [Background] Zargham-Boroujeni A, Elsagh A, Mohammadizadeh M. The Effects of Massage and Breastfeeding on Response to Venipuncture Pain among Hospitalized Neonates. Iran J Nurs Midwifery Res. 2017 Jul-Aug;22(4):308-312. doi: 10.4103/ijnmr.IJNMR_119_13. PMID 28904545
- [Result] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Result] Cong X, Ludington-Hoe SM, McCain G, Fu P. Kangaroo Care modifies preterm infant heart rate variability in response to heel stick pain: pilot study. Early Hum Dev. 2009 Sep;85(9):561-7. doi: 10.1016/j.earlhumdev.2009.05.012. Epub 2009 Jun 7. PMID 19505775
- [Result] Erkut Z, Yildiz S. The Effect of Swaddling on Pain, Vital Signs, and Crying Duration during Heel Lance in Newborns. Pain Manag Nurs. 2017 Oct;18(5):328-336. doi: 10.1016/j.pmn.2017.05.007. Epub 2017 Aug 2. PMID 28779961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: All neonates who was delivered to the hands crochet octopus during data collection process
- Control Group: All neonates who was not delivered to the hands crochet octopus during data collection process
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Median (Inter-Quartile Range); unit: days]
  Neonate's Age (day) | 8 [6 to 10] | 8 [6 to 10] | 8 [6 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 20 | 23 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 50 | 50 | 100
Neonatal Infant Pain Score [Median (Inter-Quartile Range); unit: scale score] — It is a 6-itemed scale developed to assess the pain occuring due to interventions implemented to term and premature infants. The scoring of the scale was realized by assessing five behavioral classification (mimics, crying, movements of arms and legs, wakefulness state) and one physological parameter (type of respiration). It needs too much time and is difficult to assess intubated infants. It is suitable for painful conditions of non-intubated infants. The lowest score of the scale is 0; the highest one is 7 and 3+ score shows the presence of pain.
  scale score | 0 [0 to 1] | 1 [0 to 1] | 0 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Neonate Infant Pain Scale Score
Description: Neonate Infant Pain Scale score calculated before, durring and after heel lance procedure whom neonates delivered crochet octopus and not delivered crochet octopus. It is a 6-itemed scale developed to assess the pain occuring due to interventions implemented to term and premature infants. The scoring of the scale was realized by assessing five behavioral classification (mimics, crying, movements of arms and legs, wakefulness state) and one physological parameter (type of respiration). It needs too much time and is difficult to assess intubated infants. It is suitable for painful conditions of non-intubated infants . Total score calculated. The lowest score of the scale is 0; the highest one is 7 and 3+ score shows the presence of pain.
Time Frame: Before the procedure (0th minute), during the procedure, after the procedure (2nd and 10th minutes)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Before procedure (0th min.) | 0 [0 to 1] | 1 [0 to 1]
  During procedure | 4 [3 to 5] | 4 [3 to 5]
  After procedure (2nd min) | 0 [0 to 1.25] | 2 [1 to 3]
  After procedure (10th min) | 0 [0 to 0] | 1 [0 to 1]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Equivalence — Power analysis was performed after the completion of the study. 98% power was obtained; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of Crying
Description: Duration of crying counted before, durring and after heel lance procedure whom neonates delivered crochet octopus and not delivered crochet octopus.
Time Frame: Before the procedure (0th minute), during the procedure, after the procedure (2nd and 10th minutes)
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 50 | 50
second
  Before procedure (0th min.) | 0 [0 to 0] | 10 [0 to 32.50]
  During procedure | 55 [31.50 to 80.25] | 60.50 [53 to 91]
  After procedure (2nd min) | 0 [0 to 20] | 33 [15 to 60]
  After procedure (10 th min) | 0 [0 to 0] | 0 [0 to 23.50]

ADVERSE EVENTS:
Time Frame: No adverse event data were collected
Description: According to the literature heel lance procedure has not serious adverse events and mortality rate
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04560374/Prot_SAP_000.pdf